CLINICAL TRIAL: NCT00455403
Title: Genotoxic Stress, Atherosclerosis, and Metabolic Syndrome- Aim 3
Brief Title: Atheroma Reduction With Chloroquine in Patients With the Metabolic Syndrome (ARCH-MS)
Acronym: ARCH-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Singulex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201110238(3); P50HL083762 (NIH)
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Metabolic Syndrome X; Overweight; Hypertension; Dyslipidemias; Prediabetic State
Keywords: Metabolic Syndrome; Atherosclerosis
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Hypertension; Dyslipidemias; Prediabetic State; Atherosclerosis | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chloroquine Subjects (Experimental): Participants will receive 80 mg of chloroquine on a daily basis.
  Interventions: Drug: Chloroquine
- Placebo Subjects (Placebo Comparator): Participants will receive a placebo comparator tablet on a daily basis.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Chloroquine — One tablet of 80 mg of chloroquine on a daily basis for 12 months followed by 12 months off drug with 1 visit at month 24
  Other Names: Arlen
  Arms: Chloroquine Subjects
Drug: Placebo Comparator — Chloroquine Placebo tablet daily for 12 months followed by 12 months off drug with 1 visit at month 24
  Other Names: placebo
  Arms: Placebo Subjects

SUMMARY:
Metabolic syndrome consists of a group of co-occuring conditions that increase an individual's risk of developing heart disease, stroke, and diabetes. The purpose of this study is to evaluate the long-term effectiveness of chloroquine, a protein-activation medication, at reducing the progression of atherosclerosis in patients with the metabolic syndrome.

Sub-study: Vascular endothelial growth factor(VEGF)and Cardiometabolic Risk, The purpose is to determine if the association of VEGF with atherosclerosis indicates that it should be a marker of the disorder.

DETAILED DESCRIPTION:
Metabolic syndrome is one of the most common disorders in industrialized countries. It consists of abnormal serum lipids, glucose intolerance, elevated blood pressure, and central obesity in the setting of insulin resistance. The syndrome substantially increases the risk of developing diabetes and vascular disease, but there is no clear unifying approach to treat this disorder. In animals, activation of the protein ataxia telangiectasia mutated (ATM) using the antimalarial drug chloroquine improves features of metabolic syndrome and decreases atherosclerosis, a build-up of fatty plaque within arteries. The purpose of this study is to examine the effect of long-term treatment with low doses of chloroquine on atherosclerosis in people with metabolic syndrome.

At a baseline study visit, participants will undergo an ultrasound of the neck to evaluate carotid artery intima-media thickness (IMT) and MRI to evaluate plaque composition. In addition, blood will be collected for laboratory testing and blood pressure will be measured. Participants will then be randomly assigned to receive either placebo or chloroquine. Study visits will occur every 3 months for 1 year. At each visit, blood pressure will be measured and blood will be collected. At Months 6 and 12, a repeat ultrasound will be performed. At month 12 a repeat carotid MRI is performed. Participants will attend one follow-up visit at Month 24 and will undergo a final ultrasound.

Sub-Study: VEGF and Cardiometabolic Risk, (This is an observational, case-study of existing baseline plasma and carotid intimal-medial thickness measurements) VEGF is also closely linked to vascular disease. From cell culture and animal models it is known that VEGF is increased in atherosclerotic lesions. It is controversial whether that relationship is causative or reparative. Both pro- and anti-VEGF therapies have been proposed for atherosclerosis. However, the association of VEGF with atherosclerosis indicates that it should be a marker of the disorder, which is the hypothesis we wish to test. No previous studies of circulating VEGF have been published.

Other markers may be related to vascular disease or VEGF in this dataset. Tumor necrosis factor (TNF)-alpha results in increased expression of VEGF and may be correlated positively with VEGF. By Erenna Technology testing, cardiac troponin I can be measured at levels much lower than current clinical assays and is expected to be elevated in ischemia but not necessarily in the stable vascular disease anticipated in our subjects. High sensitivity C-reactive protein (hsCRP)has been proposed as a marker for vascular disease that merits drug treatment in its own right and may also be correlated with VEGF and vascular disease. However, currently the relationship between hsCRP and vascular disease is not completely clear.

For this preliminary VEGF study observational data from the baseline only will be studied. Baseline testing includes carotid artery intimal-medial thickness, carotid MRI, lipid panel, complete blood count, comprehensive metabolic chemistry panel, Thyroid-stimulating hormone (TSH) and glucose tolerance test with plasma insulin and glucose responses. Plasma collected at baseline (approximately 1 ml) will be transferred to Singulex on dry ice. Samples will be coded but will not contain patient identifiers. Erenna Technology assays will be done for VEGF-A, cardiac troponin I,TNF-alpha, interleukin-6, interleukin-17A, and other cytokines at Singulex. This method utilizes single-photon counting of visible light to improve assay sensitivity. Separately, Washington University's Core Lab for Clinical Studies (CLCS) will determine hsCRP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metabolic syndrome, as determined by at least three of the following five criteria:

  1. Elevated fasting triglyceride level greater than 150 mg/dL
  2. Low HDL cholesterol levels: less than 50 mg/dL for women and less than 40 mg/dL for men
  3. Hypertension (greater than or equal to 130/85 mm Hg and less than or equal to 160/100 mm Hg) untreated; or hypertension controlled (less than or equal to 150/90 mm Hg) on a stable medication regimen for 4 weeks prior to baseline visit.
  4. Increased waist circumference: greater than 35 inches in women and greater than 40 inches in men
  5. Elevated fasting glucose level greater than or equal to 100 mg/dL and less than or equal to 126 mg/dL
* Willing to use acceptable form of birth control
* Subjects may be on a stable doses of a statin drug for at least 3 months
* Subjects may be on a stable doses of L-thyroxine for at least 3 months

Exclusion Criteria:

* Prior travel treatment with chloroquine or hydroxychloroquine as follows:

  1. Any exposure in the past 2 years
  2. More than 30 days of therapy if exposure was between 2 and 5 years ago
  3. More than 90 days of therapy if exposure was between 5 and 10 years ago
  4. More than 6 months of therapy if exposure was 10 to 20 years ago
  5. More than 1 year of therapy if exposure was 20 to 30 years ago
  6. No limit if last exposure was more than 30 years ago (e.g., during the Vietnam conflict)
* Morbid obesity (body mass index [BMI] greater than 45)
* Coronary artery disease or other vascular disease
* History of stroke
* Significant kidney disease (estimated glomerular filtration rate (eGFR)less than 60 mL/min/1.73 m2)
* Diabetes
* Seizure disorder
* History of psoriasis
* Blood disorders, including anemia (i.e., hemoglobin levels less than 13 g/dL in men and less than 12 g/dL in women)
* Current malignancy or active treatment for recurrence prevention, example tamoxifen. Cancer considered to be cured, either as a result of surgery or other treatment is not exclusionary.
* Asthma requiring daily beta agonist therapy or intermittent oral steroids is exclusionary. Inhaled steroids are acceptable. Obstructive sleep apnea will be allowed if Continuous Positive Airway Pressure (CPAP) or other therapy has been stable for 6 months. Other active respiratory diseases are excluded.
* Liver disease, or liver function test results greater than twice the normal value
* Active infection, including HIV
* Serious illness requiring ongoing medical care or medication
* Treatment with atypical anti-psychotic medication. Treatment with any other medication for psychiatric illness, unless on a stable dose for 6 weeks prior to enrollment. Patients with unstable psychiatric disorders are excluded per the decision of the study MD regardless of medication history.
* Receiving any of the following lipid lowering medications: niacin, fibrates, or fish oils greater than 1 gram
* Uncontrolled hypertension (blood pressure greater than or equal to 150/90) at baseline visit.
* Need for daily over the counter medications, or currently taking cimetidine or greater than 1000 IU vitamin E daily and unwilling to reduce or discontinue the use of vitamin E or discontinue cimetidine for the duration of the study. Patients taking greater than 1000 IU of vitamin E should reduce the dose 30 days prior to randomization.
* Pregnant, breastfeeding, or intending to become pregnant
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Retinal disease
* Auditory disease or hearing loss; patients with total, irreversible hearing loss can be enrolled
* Participation in another clinical trial within past 30 days prior to screening and 60 days prior to randomization. Questionnaire or observational studies are not exclusionary.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay F. Semenkovich, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] McGill JB, Johnson M, Hurst S, Cade WT, Yarasheski KE, Ostlund RE, Schechtman KB, Razani B, Kastan MB, McClain DA, de las Fuentes L, Davila-Roman VG, Ory DS, Wickline SA, Semenkovich CF. Low dose chloroquine decreases insulin resistance in human metabolic syndrome but does not reduce carotid intima-media thickness. Diabetol Metab Syndr. 2019 Jul 29;11:61. doi: 10.1186/s13098-019-0456-4. eCollection 2019. PMID 31384309
- [Derived] Razani B, Feng C, Semenkovich CF. p53 is required for chloroquine-induced atheroprotection but not insulin sensitization. J Lipid Res. 2010 Jul;51(7):1738-46. doi: 10.1194/jlr.M003681. Epub 2010 Mar 5. PMID 20208057
- See also: click here for Washington University Research Participant Registry — https://vfh.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility included adults with at least 3 criteria of metabolic syndrome but who did not have diabetes. Subjects were studied in the setting of a single academic health center.
Pre-assignment Details: 241 participants screen failed
Period: Overall Study
Arm/Group | Chloroquine Subjects | Placebo Subjects
Started | 59 | 57
Completed | 56 | 51
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroquine Subjects | Placebo Subjects | Total
Number analyzed (Participants) | 59 | 57 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 53 | 104
  >=65 years | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12) | 55 (9) | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 33 | 77
  Male | 15 | 24 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Carotid Intima-media Thickness From Baseline to Year 1
Description: A noninvasive predictor of cardiovascular events, Carotid artery intima-media thickness (CIMT) was measured from B-mode images by a single sonographer using standard approaches
Time Frame: Measured at baseline and year 1
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: millmeter
Arm/Group | Chloroquine Subjects | Placebo Subjects
Number analyzed (Participants) | 59 | 57
millmeter
  Baseline | 0.766 (0.17) | 0.765 (0.13)
  Year 1 | 0.758 (0.16) | 0.768 (0.11)
Statistical Analysis 1: Comparison: Chloroquine Subjects vs Placebo Subjects; Test type: Superiority or Other; p = 0.7279, Mixed Models Analysis — Applies to row Title "year 1"; Mean Difference (Net) = 0.010 — applies to row title "year 1"

ADVERSE EVENTS:
Time Frame: 2 years 6 months
Arm/Group | Chloroquine Subjects | Placebo Subjects
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/57
Serious Adverse Events (participants affected / at risk) | 5/59 | 2/57
Other Adverse Events (participants affected / at risk) | 39/59 | 37/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroquine Subjects (N=59) | Placebo Subjects (N=57)
Prostate Cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
Right Knee Replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
transverse myelitis (Nervous system disorders) | 1 (1) | 0 (0)
carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
cutaneous staphylococcus infection (Infections and infestations) | 1 (1) | 0 (0)
acute appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
positive PPD (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroquine Subjects (N=59) | Placebo Subjects (N=57)
Infections (Infections and infestations) | 39 (51) | 37 (42)
allergy/immunology (Immune system disorders) | 5 (51) | 10 (42)
CNS (Nervous system disorders) | 5 (51) | 3 (57)
Psychiatric (Psychiatric disorders) | 5 (51) | 6 (57)
ocular (Eye disorders) | 16 (51) | 10 (57)

LIMITATIONS AND CAVEATS:
One limitation of the study is that it may have been underpowered to detect a difference in CIMT. Sample size estimates at the time of initiation of these studies were based on reports showing that insulin sensitizers had effects on CIMT with groups of 31-57 subjects, but subsequent work indicated the need for larger sample sizes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes